CLINICAL TRIAL: NCT01737684
Title: A Two-Part, Open-Label, Single-Dose Study to Investigate the Pharmacokinetics of MK-4618 in Patients With Hepatic Insufficiency
Brief Title: A Single-Dose Study of the Pharmacokinetics of Vibegron (MK-4618) in Adults With Hepatic Insufficiency (MK-4618-013)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4618-013
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Results first posted 2016-06-22 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — N-(4-((5-(hydroxy(phenyl)methyl)pyrrolidin-2-yl)methyl)phenyl)-4-oxo-4,6,7,8-tetrahydropyrrolo(1,2-a)pyrimidine-6-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Participants With Moderate Hepatic Insufficiency (Experimental): Participants with moderate hepatic insufficiency will receive a single oral dose of vibegron 100 mg.
  Interventions: Drug: Vibegron
- Healthy Matched Control Participants (Experimental): Participants who are healthy will receive a single oral dose of vibegron 100 mg.
  Interventions: Drug: Vibegron
- Participants With Mild Hepatic Insufficiency (Experimental): Participants with mild hepatic insufficiency will receive a single oral dose of vibegron 100 mg.
  Interventions: Drug: Vibegron

INTERVENTIONS:
Drug: Vibegron — 50 mg tablet, oral
  Other Names: MK-4618

SUMMARY:
This study will investigate the pharmacokinetics of a single oral dose of vibegron (MK-4618) administered to participants with moderate hepatic insufficiency and healthy participants matched for age, gender, and body mass index (BMI). Participants may be enrolled with mild hepatic insufficiency.

DETAILED DESCRIPTION:
This study is planned to be conducted in two parts. Part 1 of the study will include participants with moderate hepatic insufficiency and healthy participants. If Part 2 is conducted, Part 2 of the study will include participants with mild hepatic insufficiency.

ELIGIBILITY:
Inclusion Criteria

For both healthy participants and participants with hepatic insufficiency:

* Continuous non-smokers who haven't used nicotine-containing products for at least 3 months prior to study drug administration
* Body mass index (BMI) ≤39 kg/m^2
* Good health based on medical history, physical examination, vital signs, laboratory safety tests, and electrocardiogram (ECG)
* Females of childbearing potential must be sexually inactive for 14 days prior to study drug administration and throughout study or use acceptable birth control method
* Females of non-childbearing potential must have undergone an acceptable sterilization procedure at least 6 months prior to Day 1 of study or be postmenopausal with amenorrhea for at least 1 year prior to Day 1
* Non-vasectomized males must agree to use a condom with spermicide or abstain from sexual intercourse during the trial and for 3 months after study drug administration

For participants with hepatic insufficiency only:

* Diagnosis of chronic, stable, hepatic insufficiency
* For Part 1 Participants: Child-Pugh scale range from 7 to 9
* For Part 2 Participants: Child-Pugh scale range from 5 to 6

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-01-15 (Actual); Primary Completion 2013-06-14 (Actual); Study Completion 2013-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was planned to be conducted in two parts. Part 1 was to include participants with moderate hepatic insufficiency and healthy participants. Part 2 was to include participants with mild hepatic insufficiency. After a review of the safety and pharmacokinetic data from Part 1, a decision was made not to conduct Part 2.
Groups:
- Participants With Moderate Hepatic Insufficiency; Healthy Matched Control Participants: Participants received a single oral dose of vibegron 100 mg on Day 1.
- Participants With Mild Hepatic Insufficiencey: Participants with mild hepatic insufficiency were to receive a single oral dose of vibegron 100 mg.
Period: Overall Study
Arm/Group | Participants With Moderate Hepatic Insufficiency | Healthy Matched Control Participants | Participants With Mild Hepatic Insufficiencey
Started | 8 | 8 | 0 (Participants with mild hepatic insufficiency were not enrolled in study.)
Completed | 8 | 8 | 0 (Participants with mild hepatic insufficiency were not enrolled in study.)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All Enrolled Participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants With Moderate Hepatic Insufficiency | Healthy Matched Control Participants | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Full Range); unit: Years] | 58 [51 to 66] | 54 [45 to 60] | 56 [45 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration Time Curve From 0 to Infinity (AUC0-∞) After a Single Oral Dose of Vibegron 100 mg
Description: Blood samples were collected for determination of vibegron levels predose and at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 120, 216, and 336 hours after dosing.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 120, 216, and 336 hours postdose
Population: Per Protocol (PP) population, which included the subset of participants who complied with the protocol sufficiently to ensure that the data were likely to exhibit the effects of treatment, according to the underlying scientific model.
Measure: Geometric Mean (95% Confidence Interval); unit: uM•hr
Arm/Group | Participants With Moderate Hepatic Insufficiency | Healthy Matched Control Participants
Number analyzed (Participants) | 8 | 8
uM•hr | 4.10 [3.25 to 5.16] | 3.23 [2.56 to 4.07]
Statistical Analysis 1: Comparison: Participants With Moderate Hepatic Insufficiency vs Healthy Matched Control Participants; Test type: Superiority or Other; ANCOVA; Geometric least-squares mean ratio = 1.27, 90% CI 2-sided [0.96 to 1.67]

2. Secondary Outcome: Apparent Clearance (CL/F), Calculated as Dose/AUC0-∞, After a Single Oral Dose of Vibegron 100 mg
Description: as for outcome 1
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 120, 216, and 336 hours postdose
Population: Per Protocol (PP) population, which included participants who complied with the protocol sufficiently to ensure that the data were likely to exhibit the effects of treatment, according to the underlying scientific model.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Participants With Moderate Hepatic Insufficiency | Healthy Matched Control Participants
Number analyzed (Participants) | 8 | 8
L/hr | 56.0 (31.2) | 68.3 (36)

3. Secondary Outcome: Apparent Volume of Distribution During the Terminal Phase (Vd/F) After a Single Oral Dose of Vibegron 100 mg
Description: as for outcome 1
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 120, 216, and 336 hours postdose
Population: PP population, which included participants who complied with the protocol sufficiently to ensure that the data were likely to exhibit the effects of treatment, according to the underlying scientific model.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Participants With Moderate Hepatic Insufficiency | Healthy Matched Control Participants
Number analyzed (Participants) | 8 | 8
L | 7640 (33.3) | 9120 (30.7)

4. Secondary Outcome: Maximum Observed Plasma Drug Concentration (Cmax) After a Single Oral Dose of Vibegron 100 mg
Description: as for outcome 1
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 120, 216, and 336 hours postdose
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Arm/Group | Participants With Moderate Hepatic Insufficiency | Healthy Matched Control Participants
Number analyzed (Participants) | 8 | 8
nM | 378 [265 to 540] | 281 [197 to 401]
Statistical Analysis 1: Comparison: Participants With Moderate Hepatic Insufficiency vs Healthy Matched Control Participants; Test type: Superiority or Other; ANCOVA; Geometric least-squares mean ratio = 1.35, 90% CI 2-sided [0.88 to 2.06]

5. Secondary Outcome: Time to Maximum Observed Plasma Drug Concentration (Tmax) After a Single Oral Dose of Vibegron 100 mg
Description: as for outcome 1
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 120, 216, and 336 hours postdose
Population: as for outcome 3
Measure: Median (Full Range); unit: hr
Arm/Group | Participants With Moderate Hepatic Insufficiency | Healthy Matched Control Participants
Number analyzed (Participants) | 8 | 8
hr | 1.00 [0.50 to 3.00] | 1.50 [0.50 to 4.00]

6. Secondary Outcome: Apparent Terminal Half-life (t½) After a Single Oral Dose of Vibegron 100 mg
Description: as for outcome 1
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 120, 216, and 336 hours postdose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Participants With Moderate Hepatic Insufficiency | Healthy Matched Control Participants
Number analyzed (Participants) | 8 | 8
hr | 94.54 (8.88) | 92.48 (9.37)

ADVERSE EVENTS:
Time Frame: Up to 336 hours post-dose
Description: The All Subjects as Treated (AST) population, which consisted of all participants who received at least 1 dose of the investigational drug, was used for the safety analysis.
Arm/Group | Participants With Moderate Hepatic Insufficiency | Healthy Matched Control Participants
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 1/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Moderate Hepatic Insufficiency (N=8) | Healthy Matched Control Participants (N=8)
Flushing (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication or presentation.